CLINICAL TRIAL: NCT03383419
Title: Transplant of Redeemed Organs by Judicious Administration of New Direct-Acting Antivirals for Hepatitis-C Heart Recipients
Acronym: TROJAN-C
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 018-009
Record Dates: First submitted 2017-12-07; First posted 2017-12-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure
Keywords: Heart Failure, Heart Transplant
MeSH Terms: conditions — Heart Failure | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Epclusa® will be started within 14 days of quantifiable viremia and continued for 12 weeks. Within 24 hours prior to first-dose of treatment, HCV genotype will be sent from transplant recipient.
  Interventions: Drug: Epclusa

INTERVENTIONS:
Drug: Epclusa — If and when these recipients develop confirmed viremia by HCV PCR, Epclusa® therapy will be administered for a 12-week course.

SUMMARY:
This phase II, multi-center, open-label study will evaluate the safety and efficacy of utilizing HCV-positive donors for heart transplant in HCV-negative recipients treated with sofosbuvir 400 mg / velpatasvir 100 mg (Epclusa®).

DETAILED DESCRIPTION:
utilizing HCV-positive donors (defined as HCV-NAT positive) for heart transplantation in HCV-negative recipients treated with Epclusa®.

Subjects will be identified from the heart transplantation waitlist. Subjects who, according to the judgement of the Investigator, would have a net mortality benefit from cardiac transplantation irrespective of donor HCV status will be asked if they agree to receive a heart transplant from an HCV-positive donor. Subjects who sign consent and receive a heart transplant from an HCV-positive donor will be enrolled.

Consented subjects who do not demonstrate immunity to hepatitis B (manifest as negative qualitative or quantitative Hepatitis B surface Ab) will be encouraged to immediately begin a non-infectious recombinant hepatitis B surface antigen vaccination series, combined with, or in parallel to, an inactive hepatitis A vaccination at the treating clinician's discretion.

Enrolled recipients will be closely surveilled with serial HCV polymerase chain reaction (PCR) as inpatients during the immediate post-OHT hospitalization and subsequently as specified in the post-transplant period assessements. Donor serum will be collected at transplant harvest and will be sent by the transplant center for HCV NAT and genotyping. If and when these recipients develop confirmed viremia by HCV PCR, Epclusa® therapy will be administered for a 12-week course. The study drug, Epclusa®, will be provided by Gilead Sciences, Inc. Study drug, Epclusa®, comes in bottles that contain 28 tablets each. Serologic data will also be collected. If an enrolled subject does not develop quantifiable viremia by week 12, they will be followed by standard of care surveillance, with additional standard of care surveillance per UNOS mandate for CDC-increased-risk donors and discontinued from study; additional subjects may be enrolled at the Principal Consortium Investigator's discretion to complete 20 Epclusa®-treated subjects according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and capable of providing written informed consent
2. Age ≥ 18 years
3. Listed for isolated orthotopic heart transplant
4. HCV seronegative (or, if HCV seropositive, then subject must be PCR negative on at least 2 draws consistent with a spontaneously cleared or fully-treated and cleared prior infection; in this case last anti-HCV antiviral dose must be ≥12 weeks ago and 2 negative titers ≥12 weeks after completion of the antiviral regimen)

Exclusion Criteria:

1. Listed for combined organ transplant
2. Any of the following liver disease states, including:

   1. History of HCV viremia detectable by either HCV qualitative or quantitative PCR unless deemed cured (SVR-12),
   2. Hepatitis B surface Ag positive(unless clinically determined to be previously negative and acutely positive due to vaccination with recombinant surface antigen) or detectable hepatitis B DNA,
   3. Cirrhosis, as indicated by liver biopsy,
   4. Portal hypertension as indicated by a hepatic venous pressure gradient > 5 mm Hg and/or the presence of esophageal varices e.) ALT and AST > 3x ULN unless adjudicated to be from a non-hepatic cardiac or skeletal muscle source,
3. History of prior solid organ transplant
4. Pregnant individuals
5. History of HIV infection
6. History of severe renal disease currently requiring dialysis. Chronic kidney disease with creatinine clearance <30 ml/min/1.73m2 (by MDRD method) at screening or on last two consecutive measurements before acceptance of transplant organ offer
7. Patients who have undergone or who will undergo immune desensitization therapy
8. Prospective-positive cross-match or predicted positive cross-match
9. Patients unwilling to notify their sexual partner(s) of participation in this trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-03-20 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Sustained virologic response after 12 weeks of treatment | 12 weeks
  To evaluate the number of patients with sustained virologic response (SVR) 12 weeks after discontinuation of therapy.

SECONDARY OUTCOMES:
1-year post-transplant survival | 1 year
  To evaluate the number of patients who survive 1-year post-transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Shelley A Hall, MD, FACC, FHFSA, Study Chair — Baylor University Medical Center/ Baylor Scott & White Research Institute
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Duke University Medical Center, Durham, North Carolina
  - Baylor University Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Mozaffari E, Chandak A, Zhang Z, Liang S, Thrun M, Gottlieb RL, Kuritzkes DR, Sax PE, Wohl DA, Casciano R, Hodgkins P, Haubrich R. Remdesivir Treatment in Hospitalized Patients With Coronavirus Disease 2019 (COVID-19): A Comparative Analysis of In-hospital All-cause Mortality in a Large Multicenter Observational Cohort. Clin Infect Dis. 2022 Aug 24;75(1):e450-e458. doi: 10.1093/cid/ciab875. PMID 34596223